CLINICAL TRIAL: NCT06850701
Title: The Effect of Mindfulness-Based Stress Reduction Programme on Stress, Anxiety, Self-Compassion and Prenatal Attachment in Pregnant Women With Perinatal Loss; A Randomised Controlled StudyMBSR
Brief Title: The Effect of Mindfulness-Based Stress Reduction Programme on Stress, Anxiety, Self-Compassion and Prenatal Attachment
Acronym: MBSRASPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Gul OZTAS, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KahramanmaraşSIU8
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-02

CONDITIONS: 28 Weeks of Gestation; 18 Years and Over
Keywords: perinatal loss; midwifery
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): mbsr
  Interventions: Behavioral: mbsr
- control group (Other): THERE IS NO APPLICATION OF ANY KIND
  Interventions: Behavioral: mbsr

INTERVENTIONS:
Behavioral: mbsr — In order to evaluate the effect of MBSR programme on stress, anxiety, self-compassion and prenatal attachment of pregnant women with perinatal pregnancy loss, MBSR will be applied for four weeks (two sessions per week) for a total of eight sessions in the experimental group. The intervention protocol of this study includes the entire MBSR programme consisting of two sessions per week for 1 month and homework assignments given throughout the programme. In all sessions, mindfulness exercises such as 3-minute breathing, body and breathing exercises, body scanning meditation, sitting meditation, mountain meditation, compassion meditation will be applied to the participants under the guidance of the researcher (H.G.Ö) who is trained and certified in the field of MBSR. It will be done in sessions and individual practices in an environment where pregnant women will not be disturbed at any time of the day. The live online MBSR programme will be provided through mobile communication tools. Sess

SUMMARY:
This research will be conducted to examine the effects of a mindfulness-based stress reduction (MBSR) programme on stress, anxiety, self-compassion and prenatal attachment in pregnant women with perinatal loss.

This randomised controlled trial was conducted with 80 pregnant women with perinatal loss (40 participants in the experimental group and 40 participants in the control group). The experimental group will receive a total of eight sessions of MBSR in two sessions per week for four weeks. The data of the study will be collected by Personal Information Form, Tilburg Distress in Pregnancy Scale, Self-Compassion Scale Short Form, Subjective Discomfort Unit Scale and Prenatal Maternal Attachment Scale.

DETAILED DESCRIPTION:
Perinatal loss is defined as miscarriage, stillbirth and neonatal death occurring in the first 28 days after birth ( Cassidy et al., 2018; Alvarez-Calle., & Chaves, 2023; Donegan et al. 2023). According to the World Health Organisation report, 2.6 million perinatal losses and 2.7 million neonatal deaths occurred in 2017 (WHO, 2018). Perinatal loss creates significant psychological effects for many women and in some cases can be severe enough to cause psychiatric disorders (Herbert et al., 2022). It is known that women who experience perinatal loss are more likely to experience negative mental health problems such as anxiety, stress, guilt and emotional loneliness when they become pregnant again (Cassaday ,2018; Hunter et al. 2017). Stress during pregnancy can lead to various physical consequences such as premature birth, low birth weight, gestational hypertension and increased risk of asthma (Glover, 2014; Dağlar, & Hotun Şahin, 2021).

Another important concept that reduces pregnancy stress level is self-compassion. Self-compassion helps the individual to be kinder to himself/herself and to look at himself/herself less critically (Neff, 2003). As the level of self-compassion increases, positive psychological characteristics such as psychological well-being, positive affect, life satisfaction and forgiveness increase (Bacanlı & Çarkıt, 2020). It is stated that individuals with high levels of self-compassion exhibit a more supportive and compassionate approach towards themselves, can look at events from a holistic perspective and cope with difficulties in a healthier way (Bacanlı & Çarkıt, 2020; Neff, 2023). Self-compassion also contributes to mothers' adoption of maternal roles and strengthening mother-infant attachment (Kordi & Mohamadirizi, 2018). It is stated that women who experience perinatal loss experience intense anxiety and fear of losing their baby in subsequent pregnancies, which may result in difficulties in prenatal attachment (Yılmaz, 2013). Prenatal attachment refers to the emotional bond that the mother develops with her baby throughout her pregnancy and begins to form from the early stages of pregnancy (Topaç Tuncel & Kahyaoğlu Süt, 2019).

In order to protect the general health of women, it is of great importance to evaluate the levels of stress, anxiety and depression and to implement supportive interventions when necessary. In this context, one of the non-pharmacological interventions is the mindfulness-based stress reduction (MBSR) programme (Nasrollahi et al., 2022). The MBSR programme includes training materials as well as practice sessions of four basic meditation techniques including sitting meditation, body scanning, yoga and walking meditation (Zhang et al., 2019). However, it is an eight-week programme consisting of various holistic techniques and therapeutic approaches that support the integration of mindfulness into daily life, including stress coping processes (Creswell, 2017). In the literature, it has been emphasised that the MBSR programme reduces the stress and anxiety levels of pregnant women and is effective on prenatal attachment in pregnant women (Akça et al, 2023; Gheibi et al, 2020; Feli et al, 2024). There is increasing evidence that mindfulness practice through MBSR increases self-compassion (Jiménez-Gómez et al.2022; .Birnie et al.2010; Robins et al.2012). Various intervention programmes are needed to support women's psychological well-being and to reduce stress, anxiety and depression levels during pregnancy after perinatal loss. MBSR, which is among the non-pharmacological approaches, stands out as an effective intervention method in this process (Nasrollahi et al., 2022). The MBSR programme is an eight-week training programme that includes various mindfulness techniques such as sitting meditation, body scanning, yoga and walking meditation (Zhang et al., 2019; Creswell, 2017). In the literature, it is emphasised that the MBSR programme reduces stress and anxiety in pregnant women and has positive effects on prenatal attachment (Akça et al., 2023; Gheibi et al., 2020; Feli et al., 2024). In addition, there is increasing evidence that mindfulness-based practices increase self-compassion (Jiménez-Gómez et al., 2022; Birnie et al., 2010; Robins et al., 2012).

This study was conducted as a randomised controlled trial to examine the effects of MBSR programme on stress, anxiety, self-compassion and prenatal attachment in pregnant women who experienced perinatal loss. The findings of the study are expected to contribute to the development of effective interventions that support women's psychological resilience during pregnancy after perinatal loss. As a result, this study will provide important evidence on how midwifery care services can be improved, how the need for psychosocial support can be met and how mindfulness-based approaches can be integrated into midwifery care during pregnancy after perinatal loss. Thus, by increasing the capacity of midwives to provide women-centred care, women will be supported to have a physically and psychologically healthy pregnancy process.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were between 10-28 weeks of gestation,
* had a prenatal diagnosis of pregnancy,

Exclusion Criteria:

* participation in mind-body practices or a different antenatal care programme during the study,
* unwillingness to participate in the sessions,

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Tilburg Distress in Pregnancy Scale | 1 month
  It was developed by Pop et al. in the Netherlands in 2011 for the diagnosis of distress in pregnancy. It was translated into Turkish by Çapık in 2013 after a Turkish validity and reliability study. The scale consists of a total of 16 items. It is 4-point Likert type. The lowest score that can be obtained from the total scale is 0 and the highest score is 48. The scale has two sub-dimensions as 'Negative affect' and 'Partner involvement'. The scale can be applied to pregnant women aged 12 weeks and above. Cronbach's alpha coefficient of the original scale was 0.78. The Cronbach's alpha coefficient of the Turkish form of the scale is 0.80 (Çapık et al. 2015).
Self-Compassion Scale Short Form (SCS-SS-S) | 1 month
  The Turkish validity and reliability of the scale developed by Neff (2003) was conducted by Yıldırım and Sarı (2018). The scale was found to have 11 items, a single dimension and a structure with complementary positive and negative components (Yıldırım & Sarı, 2018). Neff (2015) used the scale in parents of children with ASD and reported that self-compassion can play an important role in the well-being of parents of children with autism. A total score is used in the SCS-C scale. An increase in the scores obtained from the scale indicates a high level of self-compassion. The internal consistency coefficient of the scale is 0.75 (Yıldırım & Sarı, 2018) (ANNEX-10). In this study, the Cronbach Alpha internal consistency coefficient of the scale was 0.65 in the pretest and 0.66 in the posttest (Yıldırım & Sarı, 2018).
Subjective Units of Disturbance Scale (SUDS) | 1 month
  Developed by Wolpe, SUDS is used in energy therapies and assesses the individual's discomfort. The SUDS can be applied immediately before and at the end of the therapy. The score given serves as a concrete and basic point of departure regarding the condition of the individual at the beginning of the therapy and reflects the change at the end of the application. It has previously been used in energy therapy studies in our country (Dincer et al. 2023; Patterso, 2016). This scale is scored between 0 and 10, with 0 indicating no anxiety and 10 indicating high anxiety. As the number value increases, the discomfort experienced by the person becomes more severe. The numbers in the scale show the following statements (Wolpe, 1973).

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmama Universty, Kahramanmaraş Merkez, K.maraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No